CLINICAL TRIAL: NCT01846234
Title: Effect of Sodium Intake in Multiple Sclerosis Disease Activity
Brief Title: Sodium Intake in Multiple Sclerosis
Acronym: SALT
Status: Completed | Type: Observational
Sponsor: Fundación para la Lucha contra las Enfermedades Neurológicas de la Infancia (Other)
Responsible Party: Principal Investigator, Mauricio F. Farez, Research Associate, Fundación para la Lucha contra las Enfermedades Neurológicas de la Infancia
Other Study IDs: Salt; Salt-1 (Other Grant/Funding Number: FLENI)
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Salt
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MS patients: MS patients

SUMMARY:
Recently, it has been shown that salt (ClNa, sodium chloride) can modulate the differentiation of human and mouse TH17 cells. Indeed, mice feed with high sodium diet were described to develop more aggressive course of EAE (Experimental Autoimmune Encephalitis).

However, the role of sodium intake in MS has not been investigated. In this study we investigate the effect of sodium intake in Multiple Sclerosis (MS) clinical and radiological activity.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 18 and 50 years old
* Subject has diagnosis of relapsing-remitting MS according to McDonald criteria (2010)

Exclusion Criteria:

* Patient who had hyponatremia in the last 90 days

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: A total of 70 patients with relapsing-remitting MS according to McDonald criteria1 were recruited from the MS clinic at FLENI by attending neurologists. A second group of 52 relapsing-remitting MS patients was recluted later.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2010-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Exacerbation rate | 2 years
  Number of disease relapses during follow up time according to salt consumption

SECONDARY OUTCOMES:
Radiological activity | One year
  Number of new lesions in MRI

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio F Farez, MD MPH, Principal Investigator — Fundación para la Lucha contra las Enfermedades Neurológicas de la Infancia
Locations (1):
- FLENI, Buenos Aires, Argentina